CLINICAL TRIAL: NCT02827487
Title: Tramadol Versus Celecoxib in Reducing Pain Associated With IUD Insertion: A Double Blind Placebo Controlled Trial
Brief Title: Tramadol Versus Celecoxib in Reducing Pain Associated With IUD Insertion
Acronym: IUD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer of Gynecology and Obstetrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Celecoxib IUD
Record Dates: First submitted 2016-07-03; First posted 2016-07-11 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Tramadol; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tramadol (Active Comparator): Women will receive oral Tramadol 100mg (Trama®, Global Napi, Giza, Egypt) and an oral placebo similar to Celecoxib 2 hours before IUD insertion.
  Interventions: Drug: Tramadol; Drug: Placebo 2; Procedure: IUD
- Celecoxib (Active Comparator): Women will receive oral Celecoxib 200mg (Celebrex® 200, Pfizer, USA) and an oral placebo similar to Tramadol 2 hours before IUD insertion.
  Interventions: Drug: Celecoxib; Drug: Placebo 1; Procedure: IUD
- Placebo 1 (Placebo Comparator): Women will receive a placebo similar to Tramadol and a placebo similar to Celecoxib orally 2 hours before IUD insertion.
  Interventions: Drug: Placebo 1; Drug: Placebo 2; Procedure: IUD

INTERVENTIONS:
Drug: Tramadol — Women will receive Tramadol 100mg (Trama®, Global Napi, Giza, Egypt) orally 2 hours before IUD insertion.
  Arms: Tramadol
Drug: Celecoxib — Women will receive Celecoxib 200mg (Celebrex® 200, Pfizer, USA) orally 2 hours before IUD insertion.
  Arms: Celecoxib
Drug: Placebo 1 — Women will receive a placebo similar to Tramadol orally 2 hours before IUD insertion.
  Arms: Celecoxib; Placebo 1
Drug: Placebo 2 — Women will receive a placebo similar to Celecoxib orally 2 hours before IUD insertion.
  Arms: Placebo 1; Tramadol
Procedure: IUD — IUD insertion

SUMMARY:
Two hundred and ten women requesting IUD insertion will be randomly divided into three equal groups. To ensure blinding the double dummy technique will be used in which group 1 will receive Tramadol 100mg (Trama®, Global Napi, Giza, Egypt) orally in addition to a placebo similar to Celecoxib, group 2 will receive Celecoxib 200mg (Celebrex® 200, Pfizer, USA) in addition to a placebo similar to Tramadol, and group 3 will received a placebo similar to Tramadol in addition to a placebo similar to Celecoxib. All the drugs will be given 2 hour before the procedure.

After insertion of the IUD the women's pain perception will be assessed using a visual analogue scale (VAS) graduated from zero to 10 with zero corresponding to no pain and 10 corresponding to the worst possible pain.

DETAILED DESCRIPTION:
The intrauterine device (IUD) is a commonly used long-acting, effective and reversible method of contraception. IUD insertion is usually associated with a variable degree of pain. The majority of women experience mild pain or discomfort during IUD insertion, and some women may experience severe pain. Nulliparous women, women who delivered only by cesarean section and women remote from vaginal delivery are subgroups of women who experience more pain during IUD insertion. Prophylactic pharmacological interventions for management of pain associated with IUD insertion include nonsteroidal anti-inflammatory drugs (NSAIDs), opioid analgesics including Tramadol. Tramadol hydrochloride is an orally active centrally acting synthetic opioid. It is an atypical analgesic with a dual mechanism of action: serotonin and norepinephrine reuptake inhibition and modest l-opioid agonist. It has a lower incidence of respiratory depression, cardiac depression, side effects on smooth muscle and abuse potential as compared to typical opioid agents. Cervical ripening with prostaglandins was suggested facilitate the introduction of the IUD through the cervix, although at the cost of increased pain due to uterine cramping.

The study objective is to compare the effectiveness and side effects of oral Tramadol 100mg versus oral Celecoxib 200mg in reducing pain associated with operative outpatient hysteroscopy in an attempt to find the most effective drug with the least possible side effects to be used before IUD insertion.

Two hundred and ten women requesting IUD insertion will be randomly divided into three equal groups. To ensure blinding the double dummy technique will be used in which group 1 will receive Tramadol 100mg (Trama®, Global Napi, Giza, Egypt) orally in addition to a placebo similar to Celecoxib, group 2 will receive Celecoxib 200mg (Celebrex® 200, Pfizer, USA) in addition to a placebo similar to Tramadol, and group 3 will received a placebo similar to Tramadol in addition to a placebo similar to Celecoxib. All the drugs will be given 2 hour before the procedure. An independent person will generate the allocation sequence using computer generated random numbers.

The researchers will performed bimanual examination, introduce a speculum into the vagina and sterilized the cervix with povidone iodine before inserting the IUD according to the manufacturer recommendations.

After insertion of the IUD the women's pain perception will be assessed using a visual analogue scale (VAS) graduated from zero to 10 with zero corresponding to no pain and 10 corresponding to the worst possible pain.

Quantitative data will be statistically represented in terms of mean ± standard deviation (± SD) while categorical data will be represented as frequency and percentage. Comparison of quantitative data will be done using ANOVA test for independent samples while categorical data will be compared using Chi squared test or Fisher exact test when appropriate. A probability value (p value) less than 0.05 will be considered significant.

To the best of the investigators' knowledge this is the first trial to investigate the role of Celecoxib and oral Tramadol in reducing IUD insertion associated pain, with no previous data to calculate the sample size with. Assuming that the response will be normally distributed, the sample size is calculated to detect a mean difference of 1 unit between Tramadol and Celecoxib pain scores during the procedure (lower difference are not considered clinically relevant) using VAS assuming that the within group standard deviation will be 2. The investigators will need to study 64 cases in each group to be able to reject the null hypothesis that the population means of the Tramadol and Celecoxib are equal with probability (power) 0.8. The investigators added 6 cases to each arm accounting for any missing data and procedure failure ending in 70 cases in each group. The Type I error probability associated with this test of this null hypothesis is 0.05 using Student's t test for independent samples. Sample size calculation is done using Stats Direct statistical software version 2.7.2 for Windows, Stats Direct Ltd., Cheshire, UK.

ELIGIBILITY:
Inclusion Criteria:

* Women with expected difficult IUD insertion like nulliparous women and women with previous cesarean section.

Exclusion Criteria:

* Previous vaginal delivery.
* Submucous myoma.
* Uterine anomalies.
* Undiagnosed vaginal bleeding.
* Pelvic inflammatory disease.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain after IUD insertion | one minute after IUD insertion
  Women will mark a point corresponding to their pain on a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: AbdelGany M Hassan, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

REFERENCES:
- [Background] Hassan A, Wahba A, Haggag H. Tramadol versus Celecoxib for reducing pain associated with outpatient hysteroscopy: a randomized double-blind placebo-controlled trial. Hum Reprod. 2016 Jan;31(1):60-6. doi: 10.1093/humrep/dev291. Epub 2015 Nov 29. PMID 26621854
- [Background] Kass-Wolff JH, Fisher JE. Evidence-based pain management for endometrial biopsies and IUD insertions. Nurse Pract. 2014 Mar 13;39(3):43-50. doi: 10.1097/01.NPR.0000434094.19101.d1. PMID 24535311
- [Background] Scavuzzi A, Souza AS, Costa AA, Amorim MM. Misoprostol prior to inserting an intrauterine device in nulligravidas: a randomized clinical trial. Hum Reprod. 2013 Aug;28(8):2118-25. doi: 10.1093/humrep/det240. Epub 2013 Jun 5. PMID 23739219